CLINICAL TRIAL: NCT02337010
Title: Continuous Central Venous Oxygen Saturation Assisted Intraoperative Hemodynamic Management During Major Abdominal Surgery
Brief Title: Continuous Central Venous Oxygen Saturation Assisted Intraoperative Hemodynamic Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Domonkos Trásy (Other)
Responsible Party: Sponsor-Investigator, Domonkos Trásy, Ph.D. student; Department of Anaesthesiology and Intensive Therapy, Szeged University
Organization: Szeged University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CeVOX-study
Record Dates: First submitted 2015-01-06; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Major Abdominal Surgery; Perioperative Haemodynamic Monitoring; Perioperative Fluid Management; Perioperative Vasopressor Requirement; Postoperative Organ Function; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): In the control group if the mean arterial pressure fall below 60 mm Hg and the central venous pressure (CVP) is low fluid bolus is administered if the central venous pressure is in normal range vasopressor is given.
  Interventions: Device: CVP; Drug: Fluid bolus; Drug: Vasopressor
- CeVOX (Experimental): In the ScvO2 group patients receive interventions in two options: if the ScvO2 fall below 75% or more than 3% or if the mean arterial pressure fall below 60 mm Hg. In the former case the mean arterial pressure in the latter the ScvO2 values determined if tha patient received fluid or vasopressor or both.
  Interventions: Device: CeVOX; Drug: Fluid bolus; Drug: Vasopressor

INTERVENTIONS:
Device: CeVOX — Central venous saturation was continuously monitored by using a CeVOX monitor (Pulsion Medical Systems, Munich, Germany). The CeVOX probe (PV2022-37; Pulsion Medical Systems, Munich, Germany) was inserted into the internal jugular central venous catheter as described in the user's manual.
  Arms: CeVOX
Device: CVP — Central venous pressure was continuously monitored by using a central venous catheter. The probe was inserted into the internal jugular central vein as described in the user's manual.
  Arms: Control
Drug: Fluid bolus — If hypovolaemia was suspected fluid bolus was given in the form of 250 ml hydroxyethyl starch solution (HES, 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride, Voluven, Fresenius Kabi, Germany) over 15 minutes.
Drug: Vasopressor — If hypotension was present it was treated with vasopressor as 10 mcg bolus or continuous infusion of norepinephrine (Arterenol® Sanofi, Germany).

SUMMARY:
Patients who are scheduled for: elective oesophageal tumour resection, total gastrectomy, pancreas resection, major vascular, total cystectomy will be recruited.To investigate effects of central venous pressure (CVP) and central venous saturation (ScvO2) guided fluid management on intraoperative haemodynamic parameters, volume and vasopressor requirement, and postoperative organ function and postoperative inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing the following elective major abdominal surgery: oesophagectomy, total gastrectomy, radical cystectomy, aorta-bifemoral bypass or elective operation of abdominal aortic aneurysm.
* after surgery patients were admitted to our intensive care unit.

Exclusion Criteria:

* patients younger than 18 years
* chronic organ insufficiency: "Acute Physiology and Chronic Health Evaluation (APACHE) II" scoring system: New York Heart Association Class IV, chronic hypoxia or hypercapnia, chronic renal failure requiring renal replacement therapy, biopsy proven cirrhosis or portal hypertension and immunodeficiency.
* preoperative anaemia (haemoglobin<100g/L)
* coagulation abnormality
* and patients with chronic use of corticosteroids and non-steroid anti-inflammatory drugs
* patients requiring an operation due to malignant disease where the tumour then proved to be inoperable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative complications. | 28 days

SECONDARY OUTCOMES:
Difference in the perioperative fluid requirement | postoperative 48 hours
Difference in the perioperative vasopressor requirement | postoperative 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

REFERENCES:
- [Derived] Mikor A, Trasy D, Nemeth MF, Osztroluczki A, Kocsi S, Kovacs I, Demeter G, Molnar Z. Continuous central venous oxygen saturation assisted intraoperative hemodynamic management during major abdominal surgery: a randomized, controlled trial. BMC Anesthesiol. 2015 Jun 4;15:82. doi: 10.1186/s12871-015-0064-2. PMID 26041437